CLINICAL TRIAL: NCT02240069
Title: Residential Wood Smoke Interventions Improving Health in Native American Populations
Brief Title: Wood Smoke Interventions in Native American Populations
Acronym: EldersAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Curtis Noonan, Principal Investigator, Professor, University of Montana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 218-12; R01ES022583 (NIH)
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Respiratory; Disorder, Functional, Impaired; Respiratory Infection Other
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Education (Tx1) (Experimental): Education on best burn practices
  Interventions: Behavioral: Education (Tx1)
- Air Filtration Unit Treatment (Tx2) (Active Comparator): A 20" x 18" Filtrete air filtration unit (3M, St. Paul, MN) will be placed in the same room as the wood stove.
  Interventions: Device: Air Filtration Unit Treatment (Tx2)
- Placebo Intervention (Tx3) (Sham Comparator): A 20" x 18" Filtrete air filtration unit will be installed within the wood stove home. Instead of a high efficiency filter, the units will utilize a placebo filter.
  Interventions: Device: Placebo Intervention (Tx3)

INTERVENTIONS:
Behavioral: Education (Tx1) — Education on best burn practices
  Arms: Education (Tx1)
Device: Air Filtration Unit Treatment (Tx2) — A 20" x 18" Filtrete air filtration unit (3M, St. Paul, MN) will be placed in the same room as the wood stove
  Arms: Air Filtration Unit Treatment (Tx2)
Device: Placebo Intervention (Tx3) — A 20" x 18" Filtrete air filtration unit will be installed within the wood stove home. Instead of a high efficiency filter, the units will utilize a placebo filter.
  Arms: Placebo Intervention (Tx3)

SUMMARY:
A critical need exists for efficient community-based interventions aimed at reduction of environmental exposures relevant to health. Biomass smoke exposures due to residential wood heating are common among rural Native American communities, and such exposures have been associated with respiratory disease in susceptible populations. In many of these communities wood stoves are the most economic and traditionally preferred method of residential heating, but resource scarcity can result in burning of improper wood fuels and corresponding high levels of indoor particulate matter. Community-based participatory research techniques will be used to adapt intervention approaches to meet the cultural context of each participating community. At the community level, investigators will facilitate local development of a tribal agency-led wood bank program ensuring that elderly and/or persons with need have access to dry wood for heating. At the household level, investigators will use a three arm randomized placebo-controlled intervention trial to implement and assess education/outreach on best burn practices (Tx1). The content and delivery strategies of the education intervention will be adapted to each community according to stakeholder input. This educational intervention will be evaluated against an indoor air filtration unit arm (Tx2), as well as a placebo arm (Tx3, sham air filters). Tx3 will be used in comparison with the other two treatment arms to evaluate the penetration and efficacy of the community-level wood bank program. Outcomes will be evaluated with respect to changes in pulmonary function measures and respiratory symptoms and conditions among household elders. The investigators hypothesize that locally-designed education-based interventions at the community and household levels will result in efficacious and sustainable strategies for reducing personal exposures to indoor particulate matter, and lead to respiratory health improvements in elderly Native populations. This study will advance knowledge of cost-effective environmental interventions within two unique Native American communities, and inform sustainable multi-level strategies in similar communities throughout the US to improve respiratory health among at-risk populations.

DETAILED DESCRIPTION:
Rural Native American (NA) communities experience disproportionate disease burden compared to other US populations, with poor indoor air quality resulting from in-home biomass smoke exposures (residential wood stoves) a likely contributor to these health burden discrepancies. Epidemiological studies support the etiological association between indoor biomass smoke exposure and several domains of global disease burden, particularly with respect to pediatric respiratory tract infections and adult chronic obstructive pulmonary disease (COPD) and chronic bronchitis. Elderly populations are particularly susceptible to chronic respiratory conditions, and declining pulmonary function is associated with increased morbidity and mortality. Randomized trials in developing countries have demonstrated the impact that improved cookstove technologies have in reducing biomass smoke exposures and children's risk of acute respiratory infection. However limited knowledge is available regarding the potential improvements in NA elderly populations following wood stove interventions.

Today, a critical need exists for efficient community-based interventions aimed at promoting healthy indoor environments in at-risk communities. Financial and logistical barriers that currently exist in rural and economically disadvantaged NA communities prohibit the implementation and sustainability of many environmental health interventions. Regarding wood stoves, qualitative input from experts and Native communities underscores the need for innovative low-cost, sustainable interventions targeting the reduction of in-home biomass smoke exposures. In this proposal, investigators will test community-level and education-based household-level strategies aimed at promoting and implementing best-burn practices to improve air quality and respiratory health in at-risk elderly populations.

This proposal represents a multidisciplinary collaboration between university and tribal stakeholders from two Native American Reservations to develop, adapt, implement, and evaluate a two-level intervention to reduce exposure to indoor biomass smoke and improve respiratory health among elderly tribal members. Community-based participatory research techniques will be used to adapt intervention approaches to meet the cultural context of each participating community. At the community level, investigators will facilitate local development of tribal agency-led wood yard and distribution programs ensuring that elderly and/or persons with need have access to dry wood for heating. With community advisory guidance, investigators will use a three arm randomized placebo-controlled intervention trial to implement and assess education on best burn practices (Tx1) at the household level. This educational intervention will be evaluated against an indoor air filtration unit arm (Tx2), as well as a placebo arm (Tx3, sham air filters). Tx3 will be used in comparison with the other two treatment arms to evaluate the penetration and efficacy of the community-level fuel program. Outcomes will be evaluated with respect to changes in markers of respiratory health among elders and changes in indoor air quality (PM2.5). The investigators hypothesize that locally-designed education-based interventions, in the context of a community-based strategy focused on wood fuels, will result in efficacious and sustainable strategies for reducing personal exposures to indoor biomass smoke PM2.5 and lead to respiratory health improvements in elderly NA populations.

Specific Aims are as follows:

Aim 1. Facilitate the tribally-centered development, adaption, implementation, and evaluation of community-level wood yard and distribution programs for participating tribal households.

Aim 2. Facilitate the development, adaptation, implementation, and evaluation of household-level education strategies targeting best-burn practices (Tx1) for each participating tribal community.

Aim 3. Compare effectiveness, both within and between communities, of household-level interventions among elderly adults participating in a three-arm randomized placebo-controlled trial.

Aim 3a. Compare group changes in pulmonary function and respiratory symptoms and infections.

Aim 3b. Compare group changes in indoor and personal PM2.5 exposures.

Aim 4. Evaluate penetration, acceptance, and sustainability of community- and household-level strategies using both qualitative and quantitative data generated in collaboration with tribal community advisory boards and research participants.

Impact. The long-term goal of this project will be to reduce mortality and morbidity in NA communities from exposures related to residential home heating. This study will advance knowledge of effective interventions within two unique NA Reservations and describe improvements in sub-clinical indicators of pulmonary health in susceptible elderly populations. Reducing in-home wood smoke exposures through community level facilitation of access to proper fuels and introduction of sustainable, culturally appropriate best-burn practices will inform strategies for translation to other NA communities or similar rural and underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Tribal member from one of the two study regions
* Age 55 years or older.
* Utilize a wood stove as the primary heating source.
* Capable and willing to record symptom data and wood stove usage data, as well as complete pulmonary function testing (i.e., spirometry).

Exclusion Criteria:

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis W Noonan, Ph.D., Principal Investigator — University of Montana; Annie Belcourt, Ph.D., Principal Investigator — University of Montana; Tony J Ward, Ph.D., Principal Investigator — University of Montana
Locations (1):
- University of Montana, Missoula, Montana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this pre/post study recruited and consented participants completed baseline measures during a pre-intervention period (n=149). Randomization to arms occurred after the first (baseline) period and before the second (post-intervention) period. Six participants dropped out of the study before the randomization process. Thus, only 143 participants were randomized to a treatment arm.
Units Other Than Participants: Household
Period: Overall Study
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Started | 49; 47 Household | 47; 46 Household | 47; 45 Household
Completed | 44; 43 Household | 42; 41 Household | 45; 43 Household
Not Completed | 5; 4 Household | 5; 5 Household | 2; 2 Household
Not completed — Withdrawal by Subject | 5 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3) | Total
Number analyzed (Participants) | 49 | 47 | 47 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Specific age for one participant not disclosed; all participants 55 years or older
  years
    number analyzed (Participants) | 49 | 47 | 46 | 142
    (all) | 69.8 (9.3) | 69.8 (9.5) | 68.9 (8.7) | 69.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 31 | 100
  Male | 13 | 14 | 16 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 5
  Not Hispanic or Latino | 46 | 46 | 46 | 138
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 48 | 43 | 47 | 138
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 1 | 3 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] — Population: Valid spirometry measures captured for 133 of 143 participants
  liters
    number analyzed (Participants) | 45 | 44 | 44 | 133
    (all) | 2.1 (0.7) | 2.1 (0.6) | 2.0 (0.8) | 2.0 (0.7)
Forced vital capacity (FVC) [Mean (Standard Deviation); unit: liters] — Population: Valid spirometry measures captured for 133 of 143 participants
  liters
    number analyzed (Participants) | 45 | 44 | 44 | 133
    (all) | 2.6 (0.8) | 2.6 (0.7) | 2.5 (0.9) | 2.6 (0.8)
FEV1/FVC [Mean (Standard Deviation); unit: ratio] — Population: Valid spirometry measures captured for 133 of 143 participants
  ratio
    number analyzed (Participants) | 45 | 44 | 44 | 133
    (all) | 0.79 (0.08) | 0.80 (0.07) | 0.79 (0.08) | 0.79 (0.08)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Valid blood pressure measures captured for 130 of 143 participants
  mmHg
    number analyzed (Participants) | 42 | 45 | 43 | 130
    (all) | 132 (18) | 143 (19) | 137 (20) | 137 (19)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Valid blood pressure measures captured for 130 of 143 participants
  mmHg
    number analyzed (Participants) | 42 | 45 | 43 | 130
    (all) | 74 (11) | 79 (10) | 77 (14) | 77 (12)

OUTCOME MEASURES:

1. Primary Outcome: Post-intervention FEV1
Description: Mean of up to two post-intervention measures of forced expiratory volume at one second (FEV1), liters
Time Frame: Each participant was followed during a pre-intervention baseline (Winter 1) and a post-intervention follow-up period (Winter 2). Health measures were collected at two visits during both winter periods with each visit separated by at least three weeks.
Population: Valid post-intervention spirometry measures captured for 127 of 143 participants
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Number analyzed (Participants) | 43 | 40 | 44
liters | 1.9 (0.7) | 2.1 (0.6) | 2.0 (0.6)
Statistical Analysis 1: Comparison: Education (Tx1) vs Placebo Intervention (Tx3); Pre- to post-intervention change in FEV1 for Education group relative to Placebo group; Test type: Superiority; p = 0.10, Mixed Models Analysis; Linear mixed models with a fixed term for mean pre-intervention response measure, and a nested random effect to account for repeated measures; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.24 to 0.02]
Statistical Analysis 2: Comparison: Air Filtration Unit Treatment (Tx2) vs Placebo Intervention (Tx3); Pre- to post-intervention change in FEV1 for Filtration group relative to Placebo group; Test type: Superiority; p = 0.90, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.11 to 0.13]

2. Primary Outcome: Post-intervention FVC
Description: Mean of up to two post-intervention measures of forced vital capacity (FVC), liters
Time Frame: as for outcome 1
Population: Valid post-intervention spirometry measures captured for 127 of 143 participants
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Number analyzed (Participants) | 43 | 40 | 44
liters | 2.4 (0.7) | 2.7 (0.7) | 2.5 (0.7)
Statistical Analysis 1: Comparison: Education (Tx1) vs Placebo Intervention (Tx3); Pre- to post-intervention change in FVC for Education group relative to Placebo group; Test type: Superiority; p = 0.28, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.24 to 0.07]
Statistical Analysis 2: Comparison: Air Filtration Unit Treatment (Tx2) vs Placebo Intervention (Tx3); Pre- to post-intervention change in FVC for Filter group relative to Placebo group; Test type: Superiority; p = 0.89, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.14 to 0.16]

3. Primary Outcome: Post-intervention FEV1/FVC Ratio
Description: Mean of up to two post-intervention measures of forced expiratory volume at one second (FEV1) / forced vital capacity (FVC)
Time Frame: as for outcome 1
Population: Valid post-intervention spirometry measures captured for 127 of 143 participants
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Number analyzed (Participants) | 43 | 40 | 44
ratio | 0.78 (0.08) | 0.79 (0.08) | 0.80 (0.08)
Statistical Analysis 1: Comparison: Education (Tx1) vs Placebo Intervention (Tx3); Pre- to post-intervention change in FEV1/FVC for Education group relative to Placebo group; Test type: Superiority; p = 0.06, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.05 to 0.00]
Statistical Analysis 2: Comparison: Air Filtration Unit Treatment (Tx2) vs Placebo Intervention (Tx3); Pre- to post-intervention change in FEV1/FVC for Filter group relative to Placebo group; Test type: Superiority; p = 0.71, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.03 to 0.02]

4. Primary Outcome: Post-intervention Systolic Blood Pressure
Description: Mean of up to two post-intervention measures of systolic blood pressure, millimeters of mercury (mmHg)
Time Frame: as for outcome 1
Population: Valid post-intervention blood pressure measures captured for 128 of 143 participants
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Number analyzed (Participants) | 42 | 41 | 45
millimeters of mercury (mmHg) | 132 (16) | 139 (17) | 136 (22)
Statistical Analysis 1: Comparison: Education (Tx1) vs Placebo Intervention (Tx3); Pre- to post-intervention change in systolic blood pressure for Education group relative to Placebo group; Test type: Superiority; p = 0.39, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -3.46, 95% CI 2-sided [-11.45 to 4.54]
Statistical Analysis 2: Comparison: Air Filtration Unit Treatment (Tx2) vs Placebo Intervention (Tx3); Pre- to post-intervention change in systolic blood pressure for Filter group relative to Placebo group; Test type: Superiority; p = 0.95, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.25, 95% CI 2-sided [-7.73 to 8.24]

5. Primary Outcome: Post-intervention Diastolic Blood Pressure
Description: Mean of up to two post-intervention measures of diastolic blood pressure, millimeters of mercury (mmHg)
Time Frame: as for outcome 1
Population: Valid post-intervention blood pressure measures captured for 128 of 143 participants
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Number analyzed (Participants) | 42 | 41 | 45
millimeters of mercury (mmHg) | 75 (11) | 78 (11) | 76 (13)
Statistical Analysis 1: Comparison: Education (Tx1) vs Placebo Intervention (Tx3); Pre- to post-intervention change in diastolic blood pressure for Education group relative to Placebo group; Test type: Superiority; p = 0.65, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.00, 95% CI 2-sided [-5.42 to 3.42]
Statistical Analysis 2: Comparison: Air Filtration Unit Treatment (Tx2) vs Placebo Intervention (Tx3); Pre- to post-intervention change in diastolic blood pressure for Filter group relative to Placebo group; Test type: Superiority; p = 0.79, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.58, 95% CI 2-sided [-4.97 to 3.81]

6. Secondary Outcome: Post-intervention Indoor Fine Particulate Matter (PM2.5)
Description: Post-intervention average Indoor fine particulate matter (PM2.5) concentration
Time Frame: Each participant was followed during a pre-intervention baseline (Winter 1) and a post-intervention follow-up period (Winter 2). Indoor 48-hour PM2.5 average concentration was measured at two post-intervention visits separated by at least three weeks.
Population: Valid post-intervention PM2.5 measures captured for 123 of 143 households
Measure: Mean (Standard Deviation); unit: microgram/cubic meter
Units Other Than Participants: Household
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
Number analyzed (Participants) | 43 | 39 | 41
Number analyzed (Household) | 43 | 39 | 41
microgram/cubic meter | 38.8 (33.9) | 30.5 (51.5) | 41.6 (39.2)
Statistical Analysis 1: Comparison: Education (Tx1) vs Placebo Intervention (Tx3); Pre- to post-intervention change in indoor PM2.5 concentration for Education group relative to Placebo group; Test type: Superiority; p = 0.88, Mixed Models Analysis; Linear mixed models adjusted for pre-intervention PM2.5. The model includes a nested random term to account for repeated measures; Mean Difference (Net) = -2.9, 95% CI 2-sided [-33.6 to 42.0]
Statistical Analysis 2: Comparison: Air Filtration Unit Treatment (Tx2) vs Placebo Intervention (Tx3); Pre- to post-intervention change in indoor PM2.5 concentration for Filter group relative to Placebo group; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Mean Difference (Net) = -50.5, 95% CI 2-sided [-66.1 to -27.8]

ADVERSE EVENTS:
Time Frame: Two consecutive winter periods, approximately 16 months.
Arm/Group | Education (Tx1) | Air Filtration Unit Treatment (Tx2) | Placebo Intervention (Tx3)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/49 | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT02240069/Prot_SAP_000.pdf